CLINICAL TRIAL: NCT05166629
Title: Measuring the Effectiveness of Eatable Alphabet Cards as a Nutrition Education Tool in a Pediatric Weight Management Program
Brief Title: Eatable Alphabet as a Nutrition Education Tool
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Michelle Katzow, Assistant Professor of Pediatrics, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21-1152
Record Dates: First submitted 2021-12-03; First posted 2021-12-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Child Overnutrition; Child Obesity; Child Nutrition Disorders
Keywords: nutrition education; pediatric weight management; child overweight/obesity; fruit and vegetable consumption
MeSH Terms: conditions — Child Nutrition Disorders; Pediatric Obesity; Obesity

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care (Other): Usual care in the POWER Kids weight management program includes a nutrition assessment and education by a registered dietician nutritionist (RD). This includes taking a detailed dietary history, and providing individualized counseling, motivational interviewing, and nutrition education handouts/ web-based resources.
  Interventions: Behavioral: Usual Care
- Eatable Alphabet (Experimental): The intervention group will receive usual care, as described above, plus a set of Eatable Alphabet cards, which will be utilized during the visit for counseling and education, and given to the family to take home and use as they wish.
  Interventions: Behavioral: Eatable Alphabet

INTERVENTIONS:
Behavioral: Eatable Alphabet — Eatable Alphabet is a set of kitchen activity cards developed by ChopChop Family, in collaboration with the American Academy of Pediatrics, with funding from the CDC (https://www.chopchopfamily.org/eatable-alphabet/). It includes a series of alphabet cards with family-friendly recipes.
  Arms: Eatable Alphabet
Behavioral: Usual Care — Please see above description of usual care.
  Arms: Usual Care

SUMMARY:
This pilot randomized controlled trial will test the effectiveness of Eatable Alphabet cards, a child friendly nutrition education tool, on child weight and related behaviors in a clinical sample of 2 to 10-year-old children with overweight/obesity, referred to a pediatric weight management program.

DETAILED DESCRIPTION:
The goal of this research study is to determine whether the use of Eatable Alphabet cards in addition to standard weight management in a primary care setting will increase vegetable consumption. Additional outcomes that will be examined include fruit consumption, child engagement in meal selection and preparation, and clinic follow-up. If the intervention shows a significant effect in the above outcome measures, Eatable Alphabet cards can be implemented as a standard component of obesity management in primary care settings. It is hypothesized that the intervention will increase vegetable consumption, increase child engagement in meal selection and preparation, and increase clinic follow-up.

The study design is randomized control trial, in which the control group includes parent-child dyads receiving care as usual in the weight management program, including nutrition education, and the intervention group includes parent-child dyads receiving care as usual in the weight management program plus Eatable Alphabet cards in addition to typical nutrition education. All study participants will be families receiving care at the POWER Kids Weight Management Program at 410 Lakeville Road, with the child between the ages of 2 and 10 who have overweight or obesity. The primary outcome is parent reported frequency of child vegetable consumption. Secondary outcomes include: parent reported frequency of child fruit consumption, parent reported child engagement in meal selection/preparation, follow-up weight management visit attendance, and child anthropometric outcomes.

ELIGIBILITY:
Inclusion Criteria:

* New patient at Cohen Children's Medical Center POWER Kids weight management program (defined as not having been seen by the program within the past 2 years)
* Child between the ages of 2-10
* English-speaking

Exclusion Criteria:

- No appropriate caregiver available for consent.

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in parent reported child vegetable consumption (servings/day) | 1 month
  Parents will complete pre and post intervention/usual care survey measures of vegetable consumption.

SECONDARY OUTCOMES:
Change in parent reported child fruit consumption (servings/day) | 1 month
  Parents will complete pre and post intervention/usual care survey measures of fruit consumption.
Parent reported child engagement in meal selection/preparation | 1 month
  Parents will complete pre and post intervention/usual care survey measures of child engagement in meal selection/preparation.
Follow-up weight management visit attendance | 6 months
  We will determine whether the patient returned for scheduled follow-up visit via medical record review.
Change in child body mass index (BMI) z-score | 6 months
  Weight and height measured by clinical staff at the baseline visit and all subsequent visits over the next six months will be used to calculate body mass index (BMI=kg/m^2). Software will use Centers for Disease Control and Prevention (CDC) reference standards to convert BMI into a BMI z-score based on the child's age and sex. Change in BMI z-score will be defined as BMI z-score 6 months (+/- 3 months) after the intervention visit minus BMI z-score at the baseline intervention visit.
Change in weight for age (WFA) z-score | 6 months
  Weight measured by clinical staff at the baseline visit and all subsequent visits over the next six months will be used to generate weight for age (WFA) z-scores using CDC reference standards. Change in WFA z-score will be defined as WFA z-score 6 months (+/- 3 months) after the intervention visit minus WFA z-score at the baseline intervention visit.
Change in percent of the 95th percentile of BMI for age and sex | 6 months
  Weight and height measured by clinical staff at the baseline visit and all subsequent visits over the next six months will be used to calculate body mass index (BMI=kg/m^2). Software will use CDC reference standards to convert BMI into a percent of the 95th percentile for the child's age and sex. Change in percent of the 95th percentile will be defined as percent of the 95th percentile 6 months (+/- 3 months) after the intervention visit minus percent of the 95th percentile z-score at the baseline intervention visit.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle W Katzow, MD, MS, Principal Investigator — Northwell Health and Feinstein Institutes for Medical Research
Locations (1):
- Cohen Children's Medical Center, New Hyde Park, New York, United States

IPD SHARING:
Plan to Share IPD: No